CLINICAL TRIAL: NCT01446159
Title: A Phase 1b/2 Randomized Study of MEDI-573 in Combination With an Aromatase Inhibitor (AI) Versus AI Alone in Women With Metastatic Breast Cancer (MBC)
Brief Title: Study of MEDI-573 Plus Standard Endocrine Therapy for Women With Hormone-sensitive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-573-1030
Record Dates: First submitted 2011-09-12; First posted 2011-10-05 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Hormone-sensitive, HER-2 Negative Metastatic Breast Cancer
Keywords: MEDI-573, breast cancer, metastatic, aromatase inhibitor, anti-IGF
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — dusigitumab; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MEDI-573 10 mg/kg + AI (Experimental): Participants who will be enrolled in Phase 1b Cohort A of the study will receive intravenous infusion of MEDI-573 10 mg/kg on Day 1 of each 21-day cycle and AI of the investigator's choice (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573; Drug: Aromatase Inhibitor
- MEDI-573 30 mg/kg + AI (Experimental): Participants who will be enrolled in Phase 1b Cohort B of the study will receive intravenous infusion of MEDI-573 30 mg/kg on Day 1 of each 21-day cycle and AI of the investigator's choice (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573; Drug: Aromatase Inhibitor
- MEDI-573 45 mg/kg + AI (Experimental): Participants who will be enrolled in Phase 1b Cohort C and Phase 2 Arm 1 of the study will receive intravenous infusion of MEDI-573 45 mg/kg on Day 1 of each 21-day cycle and AI of the investigator's choice (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573; Drug: Aromatase Inhibitor
- Aromatase Inhibitor (Experimental): Participants who will be enrolled in Phase 2 Arm 2 of the study will receive oral AI of the investigator's choice (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: MEDI-573 — Intravenous infusion of MEDI-573 (10 or 30 or 45 mg/kg) will be administered on Day 1 of each 21-day cycle until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
  Arms: MEDI-573 10 mg/kg + AI; MEDI-573 30 mg/kg + AI; MEDI-573 45 mg/kg + AI
Drug: Aromatase Inhibitor — Aromatase inhibitor of the investigator's choice (letrozole, anastrozole, or exemestane) will be provided orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.

SUMMARY:
Study to evaluate the safety, tolerability, antitumor activity, and pharmacology of MEDI-573 in combination with an aromatase inhibitor (AI) in adult subjects with HR+, HER2-negative MBC.

DETAILED DESCRIPTION:
This is a Phase 1b/2, multicenter, open-label study to evaluate the safety, tolerability, antitumor activity, and pharmacology of MEDI-573 in combination with an AI in adult subjects with HR+, HER2-negative MBC. This study has 2 phases: a dose-evaluation phase (Phase 1b) and a randomization phase (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed MBC not deemed amenable to curative surgery or curative radiation therapy
* Tumors are positive for ER, PgR, or both
* Tumors must be negative for HER2 (by FISH, CISH or IHC)
* Female gender and age ≥ 18 years at time of study entry
* Postmenopausal
* Karnofsky Performance Status ≥ 70
* Life expectancy of ≥ 6 months

Exclusion Criteria:

* Subjects who received prior chemotherapy, hormonal therapy, immunotherapy or biologic therapy for advanced or metastatic disease with the following exceptions:

  * Prior adjuvant therapy with an AI and/or tamoxifen is allowed, provided treatment ended at least 2 weeks prior to the first dose of MEDI-573
  * Prior neoadjuvant and/or adjuvant chemotherapy for breast cancer is allowed
* Extensive symptomatic visceral disease including hepatic involvement and pulmonary lymphangitic spread of tumor, or disease that is considered by the investigator to be rapidly progressing or life threatening (eg, subjects who are intended for chemotherapy)
* Active brain metastases with the exception of subject has been treated and are asymptomatic and there has been no evidence of CNS progression for at least 4 weeks of first dose of MEDI-573
* Evidence of ongoing spinal cord compression or leptomeningeal carcinomatosis
* Unresolved toxicities from prior therapy with the exception of alopecia that have not resolved to ≤ Grade 1 at the time of starting study treatment
* Previous treatment with agents that target the IGF receptor
* History of allergy or reaction attributed to compounds of chemical or biologic composition similar to those of MEDI-573 or AI
* History of another invasive malignancy within 5 years except for curatively resected nonmelanoma skin cancer or carcinoma in situ of the cervix
* Poorly controlled diabetes mellitus

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2011-06-13 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (65):
- United States (31):
  - Research Site, Scottsdale, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Pleasant Hill, California
  - Research Site, Stamford, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Athens, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Albuquerque, New Mexico
  - Research Site, Lake Success, New York
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Richmond, Virginia
- Belgium (7):
  - Research Site, Aalst
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Mons
- Canada (3):
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
- France (2):
  - Research Site, Le Mans
  - Research Site, Montpellier
- Germany (4):
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, München
  - Research Site, Witten
- Hungary (2):
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
- Israel (6):
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Research Site, Lodz, Poland
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Nassau, The Bahamas
- United Kingdom (5):
  - Research Site, Cardiff
  - Research Site, London
  - Research Site, Southampton
  - Research Site, Stoke-on-Trent
  - Research Site, Wolverhampton

REFERENCES:
- See also: CD-ON-MEDI-573-1030-Protocol_amendment 3_redaction-PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=50&filename=CD-ON-MEDI-573-1030-Protocol_amendment%203_redaction-PDF-A.pdf
- See also: CD-ON-MEDI-573-1030-SAP-V1_and_V2_Final_Redacted_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=50&filename=CD-ON-MEDI-573-1030-SAP-V1_and_V2_Final_Redacted_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 10 countries (Belgium, Canada, France, Germany, Hungary, Israel, Spain, Poland, United Kingdom, USA).
Pre-assignment Details: A total of 187 participants were screened in the study. Of which, 183 participants were treated with study drugs.
Groups:
- MEDI-573 10 mg/kg + Aromatase Inhibitor (AI): Participants enrolled in Phase 1b of the study and received intravenous infusion of MEDI-573 10 mg/kg on Day 1 of each 21-day cycle and AI of the investigator's choice (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
- MEDI-573 30 mg/kg + AI: Participants enrolled in Phase 1 b of the study and received intravenous infusion of MEDI-573 30 mg/kg on Day 1 of each 21-day cycle and AI (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
- MEDI-573 45 mg/kg + AI: Participants received intravenous infusion of MEDI-573 45 mg/kg on Day 1 of each 21-day cycle and AI (letrozole, anastrozole, or exemestane) orally once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons. Three participants were enrolled in Phase 1b and 89 were enrolled in Phase 2 of the study.
- Aromatase Inhibitor: Participants enrolled in Phase 2 of the study and received oral AI (letrozole, anastrozole, or exemestane) once daily until unacceptable toxicity, documentation of disease progression, or withdrawal for other reasons.
Period: Overall Study
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Started | 3 | 3 | 92 | 85
Completed | 0 | 0 | 21 | 23
Not Completed | 3 | 3 | 71 | 62
Not completed — Withdrawal by Subject | 1 | 0 | 14 | 11
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Death | 2 | 3 | 43 | 36
Not completed — Other | 0 | 0 | 13 | 13

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who received any study therapy and were analysed per their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor | Total
Number analyzed (Participants) | 3 | 3 | 92 | 85 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (12.3) | 61.0 (8.7) | 63.2 (10.5) | 63.3 (11.0) | 63.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 92 | 85 | 183
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 7 | 6 | 13
  Not Hispanic or Latino | 3 | 3 | 85 | 79 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 6 | 1 | 8
  White | 2 | 3 | 84 | 82 | 171
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b and Phase 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A serious adverse event (SAE) is an AE that results in death, initial or prolonged inpatient hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or an important medical event. TEAEs and TESAEs are defined as AEs and SAEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years).
Time Frame: From the start of study treatment (Day 1) through 60 days after the last dose of treatment or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years)
Population: Safety population included all participants who received any study therapy and were analyzed per the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 3 | 3 | 92 | 85
Participants
  Any TEAEs | 3 | 3 | 90 | 82
  Any TESAEs | 2 | 0 | 21 | 16

2. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The AEs that occurred during Cycle 1 (Days 1 to 21) and were suspected of having a causal relationship to MEDI-573 and were >= Grade 3 in severity were considered as DLTs.
Time Frame: Up to Day 21 of Cycle 1
Population: Evaluable population included all participants in Phase 1b of the study, who received at least 1 full cycle of MEDI-573 and completed the safety follow-up through the DLT evaluation period (Days 1 to 21 of Cycle 1).
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

3. Primary Outcome: Phase 1b: Number of DLTs
Description: as for outcome 2
Time Frame: Up to Day 21 of Cycle 1
Population: as for outcome 2
Measure: Number; unit: DLT events
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 3
DLT events | 0 | 0 | 0

4. Primary Outcome: Phase 2: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from the randomization until the first documentation of disease progression or death due to any cause, whichever occurred first.
  The PFS was censored on the date of the last tumor assessment documenting absence of tumor progression for participants who had no documented progression and were still alive prior to data cut-off, dropout, or the initiation of alternate anticancer treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as >= 20% increase in the sum of diameters of target lesions and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of non-target lesions or a new lesion.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: The ITT population included all participants who received any study therapy and were analyzed per their randomized treatment group. Participants enrolled in Phase 2 of the study were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Months | 12.65 [8.15 to 15.54] | 11.33 [8.54 to 15.54]
Statistical Analysis 1: Comparison: MEDI-573 45 mg/kg + AI vs Aromatase Inhibitor; Test type: Superiority; p = 0.86, Log Rank; Hazard Ratio (HR) = 0.991, 95% CI 2-sided [0.689 to 1.429]

5. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Abnormal Clinical Laboratory Results Reported as TEAEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 3 | 3 | 92 | 85
Participants
  Anemia | 1 | 1 | 17 | 10
  Eosinophilia | 0 | 0 | 1 | 0
  Leukopenia | 0 | 0 | 0 | 3
  Lymphopenia | 0 | 0 | 1 | 2
  Neutropenia | 1 | 1 | 3 | 4
  Pancytopenia | 0 | 0 | 0 | 1
  Thrombocytopenia | 0 | 2 | 1 | 3
  Granulocyte count decreased | 0 | 1 | 0 | 0
  Hemoglobin decreased | 0 | 1 | 1 | 0
  Lymphocyte count decreased | 0 | 0 | 2 | 1
  Monocyte count decreased | 0 | 0 | 1 | 0
  Neutrophil count decreased | 0 | 0 | 2 | 0
  Neutrophil count increased | 0 | 0 | 1 | 0
  Platelet count decreased | 0 | 0 | 4 | 1
  White blood cell count decreased | 0 | 0 | 2 | 1
  Alanine aminotransferase increased | 2 | 0 | 8 | 4
  Aspartate aminotransferase increased | 2 | 1 | 6 | 4
  Blood albumin decreased | 0 | 0 | 1 | 0
  Blood albumin increased | 0 | 1 | 0 | 0
  Blood alkaline phosphatase increased | 0 | 1 | 5 | 5
  Blood bicarbonate decreased | 0 | 0 | 1 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 1
  Blood chloride decreased | 0 | 0 | 1 | 0
  Blood creatine increased | 0 | 1 | 1 | 0
  Blood creatinine decreased | 0 | 0 | 0 | 1
  Blood creatinine increased | 0 | 1 | 8 | 2
  Blood glucose increased | 0 | 0 | 1 | 1
  Blood lactate dehydrogenase increased | 0 | 0 | 1 | 1
  Blood magnesium decreased | 0 | 1 | 0 | 0
  Blood potassium decreased | 0 | 0 | 1 | 0
  Blood sodium decreased | 0 | 1 | 0 | 0
  Blood triglycerides increased | 0 | 0 | 1 | 2
  Blood urea increased | 0 | 0 | 1 | 0
  Blood uric acid increased | 0 | 0 | 3 | 1
  Gamma-glutamyl transferase decreased | 0 | 1 | 0 | 0
  Gamma-glutamyl transferase increased | 1 | 1 | 9 | 4
  Protein total decreased | 0 | 1 | 0 | 1
  Leukocytosis | 0 | 0 | 0 | 1
  Neutrophilia | 0 | 0 | 1 | 0

6. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: An abnormal vital signs that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 3 | 3 | 92 | 85
Participants
  Bradycardia | 1 | 0 | 1 | 1
  Palpitations | 1 | 0 | 1 | 2
  Pyrexia | 0 | 0 | 10 | 6
  Temperature intolerance | 0 | 0 | 1 | 1
  Body temperature increased | 0 | 0 | 1 | 0
  Aspiration | 0 | 0 | 1 | 0
  Dyspnoea | 2 | 0 | 18 | 14
  Hypertension | 0 | 0 | 8 | 13
  Hypotension | 1 | 0 | 1 | 0
  Orthostatic hypotension | 0 | 0 | 1 | 0

7. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Abnormal Electrocardiogram (ECG) Reported as TEAEs
Description: An abnormal ECG findings that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 3 | 3 | 92 | 85
Participants
  Sinus bradycardia | 1 | 0 | 2 | 0
  Sinus tachycardia | 0 | 0 | 0 | 1
  Supraventricular tachycardia | 0 | 0 | 0 | 2
  Tachycardia | 0 | 0 | 1 | 2
  Angina pectoris | 0 | 0 | 0 | 1
  Arrhythmia | 0 | 0 | 0 | 1
  Atrial fibrillation | 0 | 0 | 1 | 2
  Atrial flutter | 0 | 0 | 0 | 1
  Atrioventricular block first degree | 0 | 0 | 1 | 0
  Bradycardia | 1 | 0 | 1 | 1
  Cardiac failure | 0 | 0 | 1 | 0
  Cardiac valve disease | 0 | 0 | 1 | 0
  Palpitation | 1 | 0 | 1 | 2
  Ventricular extrasystoles | 0 | 0 | 1 | 0

8. Secondary Outcome: Phase 2: Number of Participants With Best Overall Tumor Response
Description: Tumor evaluation was based on RECIST v1.1 by CT or MRI scan as: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of target lesions and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of non-target lesions or a new lesion; not evaluable (NE): either no or only a subset of lesion measurements are made at an assessment.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Participants
  CR | 1 | 2
  PR | 23 | 21
  SD | 48 | 46
  PD | 15 | 12
  NE | 2 | 4

9. Secondary Outcome: Phase 2: Objective Response Rate (ORR)
Description: The ORR was defined as percentage of participants with confirmed complete response or confirmed partial response, where CR was defined as disappearance of all target and non-target lesions and no new lesions and PR was definded as >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Percentage of participants | 27.0 [18.1 to 37.4] | 27.1 [18.0 to 37.8]

10. Secondary Outcome: Phase 2: Time to Response
Description: Time to response was measured from treatment start to the first documentation of disease response and was evaluated only in participants who achieved objective response (confirmed CR or confirmed PR. The CR was defined as disappearance of all target and non-target lesions and no new lesions and PR was defined as >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Months | 4.22 [1.7 to 18.0] | 3.98 [1.9 to 16.8]

11. Secondary Outcome: Phase 2: Duration of Response (DR)
Description: Duration of response (DR) is measured from the first documentation of disease response to the first documented progressive disease and was evaluated only in participants who achieved objective response (confirmed CR or confirmed PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions and PR was defined as >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Months | 14.55 [4.5 to 58.8] | 17.18 [2.1 to 45.1]

12. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: Time to progression was measured from treatment start until the first documentation of disease progression. The PD was defined as >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of non-target lesions or a new lesion.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Months | 14.39 [8.34 to 18.69] | 11.33 [8.54 to 17.97]

13. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival (OS) was measured from treatment start until death.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Months | 39.39 [0.3 to 73.2] | 38.34 [0.3 to 51.6]

14. Secondary Outcome: Phase 2: Change in Tumor Size
Description: Mean change in tumor size is reported.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (Approximately 8 years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 89 | 85
Centimeters | -36.2 (35.8) | -26.8 (37.2)

15. Secondary Outcome: Phase 1b and Phase 2: Area Under the Serum Concentration-time Curve From Time Zero to Day 21 (AUC0-day21) of MEDI-573 for Cycle 1
Description: AUC0-day21 of MEDI-573 for Cycle 1 is reported.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: μg·day/mL
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
μg·day/mL | 1430 (867) | 4500 (725) | 7990 (1590)

16. Secondary Outcome: Phase 1b and Phase 2: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MEDI-573 for Cycle 1
Description: AUC0-info of MEDI-573 for Cycle 1 is reported.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: μg·day/mL
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
μg·day/mL | 1500 (955) | 4930 (691) | 9570 (2310)

17. Secondary Outcome: Phase 1b and Phase 2: Dose-Normalised Area Under the Serum Concentration-time Curve From Time Zero to Infinity (DN AUC0-inf) of MEDI-573 for Cycle 1
Description: DN AUC0-inf of MEDI-573 for Cycle 1 is reported.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: day·kg·μg/mL/mg
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
day·kg·μg/mL/mg | 150 (95.5) | 164 (23.0) | 213 (51.3)

18. Secondary Outcome: Phase 1b and Phase 2: Maximum Observed Serum Concentration (Cmax) of MEDI-573 for Cycle 1
Description: Cmax of MEDI-573 for Cycle 1 is reported.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
μg/mL | 269 (74.1) | 624 (210) | 1070 (253)

19. Secondary Outcome: Phase 1b and Phase 2: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI-573 for Cycle 1
Description: Tmax of MEDI-573 for Cycle 1 is reported.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
Day | 0.04 [0 to 0.09] | 0.07 [0.06 to 0.08] | 0.07 [0.03 to 0.17]

20. Secondary Outcome: Phase 1b and Phase 2: Systemic Clearance (CL) of MEDI-573 for Cycle 1
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by AUC(0-infinity).
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
mL/day/kg | 8.29 (3.86) | 6.17 (0.889) | 4.96 (1.13)

21. Secondary Outcome: Phase 1b and Phase 2: Terminal Half Life (t1/2) of MEDI-573 for Cycle 1
Description: The elimination half-life (t1/2) is the time measured for the serum concentration of MEDI-573 to decrease by 1 half to its original concentration.
Time Frame: Cycle 1 Days 1, 2, 8, 15, and 21 (Cycle 2 Day 1, pre-dose)
Population: The ITT population was considered for this analysis. Participants who received MEDI-573 were analyzed.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
Day | 4.38 (1.07) | 5.91 (2.09) | 8.45 (2.23)

22. Secondary Outcome: Phase 1b and Phase 2: Concentration of Insulin-like Growth Factor (IGF) I and IGF-II
Description: The mean concentration profiles of both IGF-I and IGF-II post administration of MEDI-573 in plasma were evaluated during treatment.
Time Frame: Baseline (Cycle1 Day1 pre-dose), end of treatment (EOT), and 60 days post last dose (Approximately 8 years)
Population: Safety population included all participants who received any study therapy and were analyzed per the treatment they actually received. Participants with free IGF concentration were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
Number analyzed (Participants) | 3 | 3 | 92 | 85
ng/mL
  Baseline: Free IGF-I Concentration: number analyzed (Participants) | 3 | 3 | 82 | 78
  Baseline: Free IGF-I Concentration | 2.57 (0.712) | 1.25 (0.635) | 3.49 (4.39) | 1.89 (1.24)
  Baseline: Free IGF-II Concentration: number analyzed (Participants) | 3 | 3 | 84 | 78
  Baseline: Free IGF-II Concentration | 3.81 (1.66) | 3.07 (0.709) | 3.01 (1.20) | 3.03 (1.12)
  EOT: Free IGF-I Concentration: number analyzed (Participants) | 2 | 2 | 40 | 38
  EOT: Free IGF-I Concentration | 0.724 (0.421) | 0.313 (0.0) | 0.346 (0.130) | 2.32 (3.64)
  EOT: Free IGF-II Concentration: number analyzed (Participants) | 2 | 2 | 40 | 38
  EOT: Free IGF-II Concentration | 0.625 (0.0) | 0.625 (0.0) | 0.641 (0.102) | 3.12 (1.22)
  60 days post last dose: Free IGF-I Concentration: number analyzed (Participants) | 1 | 2 | 21 | 22
  60 days post last dose: Free IGF-I Concentration | 1.54 (NA) — Not applicable as only one participant was evaluable for the specified time point. | 1.33 (0.3) | 1.02 (1.29) | 4.62 (8.52)
  60 days post last dose: Free IGF-II Concentration: number analyzed (Participants) | 1 | 2 | 21 | 22
  60 days post last dose: Free IGF-II Concentration | 1.49 (NA) — Not applicable as only one participant was evaluable for the specified time point. | 0.625 (0.0) | 0.984 (0.734) | 3.38 (1.51)

23. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI-573
Description: Participants With Positive ADA to MEDI-573 are reported.
Time Frame: Pre-infusion on Day 1 of each cycle, End of Treatment, Day 30, 60 and 90 post treatment (approximately 8 years)
Population: Participants who received MEDI-573 and were analyzed per the treatment they actually received were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI
Number analyzed (Participants) | 3 | 3 | 92
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the start of study treatment (Day 1) through 60 days after the last dose of treatment or until the participants started another anticancer therapy, whichever occurs first (approximately 8 years)
Description: An AE is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. An SAE is an AE that results in death, initial or prolonged inpatient hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or an important medical event.
Arm/Group | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) | MEDI-573 30 mg/kg + AI | MEDI-573 45 mg/kg + AI | Aromatase Inhibitor
All-Cause Mortality (participants affected / at risk) | 2/6 | 3/6 | 43/184 | 36/170
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 21/92 | 16/85
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 86/92 | 79/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) (N=3) | MEDI-573 30 mg/kg + AI (N=3) | MEDI-573 45 mg/kg + AI (N=92) | Aromatase Inhibitor (N=85)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-573 10 mg/kg + Aromatase Inhibitor (AI) (N=3) | MEDI-573 30 mg/kg + AI (N=3) | MEDI-573 45 mg/kg + AI (N=92) | Aromatase Inhibitor (N=85)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 30 (50) | 22 (39)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7) | 8 (13)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (8)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (11) | 4 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 14 (20) | 15 (21)
Asthenia (General disorders) | 1 (1) | 0 (0) | 19 (33) | 13 (18)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 9 (16) | 10 (20)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 9 (11) | 6 (11)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 9 (11) | 10 (13)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 6 (6)
Gamma-glutamyltransferase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (3) | 9 (41) | 4 (5)
Granulocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 6 (10) | 5 (7)
Weight increased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 7 (15) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (9) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 29 (49) | 21 (33)
Bone loss (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 9 (9) | 9 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 10 (12) | 8 (14)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 12 (15) | 11 (14)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 17 (48) | 10 (18)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (6) | 1 (1) | 3 (6) | 4 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (2) | 3 (11)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (7)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 5 (9) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (9)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1) | 21 (27) | 23 (32)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 34 (53) | 30 (46)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 3 (6) | 41 (96) | 27 (38)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 7 (9) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 26 (48) | 17 (26)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 8 (13) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 2 (7) | 1 (1) | 6 (14) | 4 (7)
Blood albumin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 5 (11) | 5 (10)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 8 (38) | 2 (2)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 19 (24) | 14 (16)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 10 (38) | 8 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (13)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (18) | 4 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 3 (16) | 4 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 28 (60) | 35 (73)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 10 (13) | 11 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 9 (10) | 10 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 14 (20) | 18 (43)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 16 (25) | 9 (12)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 13 (16) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 20 (29) | 19 (27)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 10 (13) | 8 (10)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 11 (12) | 4 (4)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 10 (12) | 13 (14)
Tachyphrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Breast haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 4 (5) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 19 (27) | 11 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 18 (21) | 14 (23)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (7) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (7) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (10) | 11 (12)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 13 (15) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (12) | 10 (15)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 13 (22) | 30 (46)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 8 (17) | 13 (24)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT01446159/Prot_000.pdf
  • Statistical Analysis Plan (2011-06-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT01446159/SAP_001.pdf